CLINICAL TRIAL: NCT06655415
Title: Family Members At INcreased-risk for Developing Inflammatory Bowel Disease (FIND-IBD)
Brief Title: Family Members At INcreased-risk for Developing Inflammatory Bowel Disease
Acronym: FIND-IBD
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Emily R. Lopes, MD, MPH, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2024P000791
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Disease (IBD); Ulcerative Colitis (UC); IBD-unclassified (IBD-U); Indeterminate Colitis; Crohn's Disease Colon; Crohn's Colitis; Crohn's Ileocolitis; Crohn's Gastritis; Crohn's Jejunitis; Crohn's Duodenitis; Crohn's Esophagitis; Ulcerative Proctitis; Ulcerative Proctosigmoiditis
Keywords: Inflammatory Bowel Disease; IBD; Ulcerative colitis; Crohn's disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood, stool, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Individuals who have a parent, sibling, or child with IBD but who do not have IBD themselves: Adult and adolescent (greater than 14 years of age) first-degree relatives (parents, siblings, or children) of patients with inflammatory bowel disease (including Crohn's disease, ulcerative colitis, or inflammatory bowel disease-unclassified/indeterminate colitis) but who do not have inflammatory bowel disease themselves.

SUMMARY:
First-degree relatives of people with inflammatory bowel disease ("IBD," including Crohn's disease and ulcerative colitis) have an increased risk for developing IBD themselves. This study will follow unaffected first-degree relatives (who do not have IBD) over time to understand if their behaviors, diet, and biomarkers for IBD can help predict who gets IBD and if IBD can be prevented in these high-risk individuals. Participants will be asked once per year to complete a questionnaire and have their blood, stool, and urine collected. The anticipated length of the study (registry) is approximately 10 years or longer. Parts of this study, such as the questionnaires and stool and urine collection, may be done from home, while other parts, such as the blood draw, will need to be done from Massachusetts General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Ability to complete all study visits and study-related procedures
* Ability to understand and complete study questionnaires
* Must have at least one first-degree relative with inflammatory bowel disease (Crohn's disease, ulcerative colitis, or IBD-unclassified)
* Age ≥ 14

Exclusion Criteria:

* Individuals with existing diagnoses of inflammatory bowel disease (ulcerative colitis, Crohn's disease, or IBD-unclassified)
* Evidence of clinical signs or symptoms of IBD, which will be identified on pre-screening interview with the study coordinator.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: First-degree relatives (FDRs) of those with IBD.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2034-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who develop inflammatory bowel disease | Through study completion (an anticipated 10 years)
  Participants will be queried annually on questionnaires for the development of inflammatory bowel disease (IBD), including Crohn's disease, ulcerative colitis, or IBD-U (self-reported outcome). Participants will then be asked for permission to obtain additional medical records, which will be reviewed by study investigators to confirm diagnosis of IBD.

CONTACTS AND LOCATIONS:
Overall Officials: Emily W Lopes, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be available upon reasonable request and per Mass General Brigham IRB guidelines as outlined in the ICF and detailed protocol.
Access Criteria: Collaborators interested in requesting data must submit a valid scientific question, include a statistical analysis plan, complete a data request form, and Data Use Agreement (DUA), which limits subsequent use to the terms of the approved request and requires that users maintain data security, and refrain from any attempts to re-identify research participants or engage in any unauthorized uses of the data.